CLINICAL TRIAL: NCT05208333
Title: Research on the Situation of Toxacara Infection and the Effectiveness of Albendazole Treatment Among Pupils Aged 3-15 Years in Ho Chi Minh City
Brief Title: The Effectiveness of Albendazole Treatment Among Infected Toxocara Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pham Ngoc Thach University of Medicine (Other)
Collaborators: Department of Science and Technology, Ho Chi Minh City, Viet Nam (Unknown)
Responsible Party: Principal Investigator, Thieu Ha Van, Lecturer at Department of Pediatrics (Pham Ngoc Thach University of Medicine), Principal Investigator, Clinical doctor at Children Hospital 2 Ho Chi Minh city, PhD, Pham Ngoc Thach University of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021020107KHCN
Record Dates: First submitted 2021-12-22; First posted 2022-01-26 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Toxocara Infection
Keywords: Toxocara; infection; children; Ho Chi Minh City; Albendazole; treatment; intervention; pupils
MeSH Terms: conditions — Toxocariasis; Infections | interventions — Albendazole; Tablets

STUDY DESIGN:
Intervention Model Description: We conducted a cross-sectional study among 960 pupils aged 3-15 years from Kindergartens, primary schools and secondary schools to describe the characracteristics, and determine the factors related to Toxocariasis infection. After that, we identified infected children from 960 children, we choose 146 infected children who are as sampling for intervention with treatment of Albendazole. Then, we evaluate the effectiveness of Albendazole treatment by follow-up these 146 infected children for 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albendazole treatment (Other): Treatment drugs: Albendazole (Zentel) tablets 200mg, Glaxo Wellcome Production France manufacturer .
  Dose: 15 mg/kg divided into 2 times/day x 5 days, orally after meals. Procedure: Distributing albedazol (Zentel) 200mg at school to parents or guardians, dose 15mg/kg divided into 2 times/day, instructions to take the medicine in full dose, at the right time after meals, for 5 days.
  Limiting reinfection: Advice on preventing reinfection Advice on preventing re-infection according to Vietnam Ministry of Health disease prevention guidelines
  Interventions: Drug: Albenza 200Mg Tablet

INTERVENTIONS:
Drug: Albenza 200Mg Tablet — Distributing albedazol (Zentel) 200mg at school to parents or guardians, dose 15mg/kg divided into 2 times/day, instructions to take the medicine in full dose, at the right time after meals, for 5 days.
  Limiting reinfection: Advice on preventing reinfection
  Other Names: Zentel

SUMMARY:
This study consists 2 phases. The first phase will conduct a cross-sectional study to determine the infection rate of Toxocariasis larvae, describe the clinical and paraclinical characteristics, identify risk factors related to Toxocariasis larva infection. The second phase will conduct an interventional study to evaluate the effectiveness and factors related to the Albendazole treatment on pupils infected with Toxocariasis larvae in Ho Chi Minh City.

DETAILED DESCRIPTION:
This study includes 2 phases below:

Phase 1: Cross-sectional study Sample population: total 960 pupils aged 3-15 years old from public kindergartens, primary schools, and secondary schools in Ho Chi Minh City.

Data collection will be conducted following stages below:

1. Explain counseling to parents/guardians and explain to children (for children > 9 years old) about Toxocariasis in dogs/cats, procedures for examination, testing, medication and follow-up. Clearly explain the benefits as well as the possible risks of participating in the study. If agreeing to participate, the parent/guardian and the child (over 9 years old) sign the commitment through a consent form.
2. Clinical examination by doctors of Pediatrics, Pham Ngoc Thach University of Medicine, seniority, prestige, practice certificates, undergraduate and postgraduate teaching at the hospital Children 2.
3. Fill in the data collection questionnaire
4. Taking blood for testing:

   * Type of test: Complete blood count (TPTTBM), AST, ALT, Urea, Creatinine, IgE, ELISA.
   * Place of implementation: At the school of the child selected for the study.
   * Performer: Senior and skilled pediatric nurse working at Children's Hospital 2, with good practice and professional certificates
   * Blood volume taken: 4ml (0.5ml for BM; 1.5ml for urea, creatinine, AST, ALT, IgE; 2ml for ELISA).
   * Preserve and transport blood samples to the laboratory of Children's Hospital 2 according to the procedure.
   * Treatment of accidents, if any, during the procedure: Equip shock-proof boxes and appropriate on-site first aid tools, treat them according to the protocol of the Ministry of Health, transfer the child to the nearest medical facility.
5. Make an appointment to announce test results and re-evaluate.
6. Nurturing children

Phase 2: Interventional study Children infected with Toxocariasis larvae were recruited from the cross-sectional survey based on the results of positive ELISA test for Toxocariasis, with or without increased BCAT and IgE, history and clinical symptoms.

Sample size was calculated based on the research results of Fernando (treatment within 3 months), about 146 children will be recruited about 146 children, intervention with Albendazole treatment on these children is sufficient.

Evaluation after intervention: Children after being diagnosed will be invited into intervention with Albendazole according to the protocol, continued to follow up after 1 month and 6 months in most cases.

* Within the scope of this topic, we evaluate the cure based on standards from the disease under the guidance of the Vietnam Ministry of Health in 2020

* Clinical symptoms decrease or disappear after treatment
* The ELISA test has decreased or returned negative antibody titers.
* The percentage of eosinophils, total IgE decreased or returned to normal values.

Data collection process includes the steps of intervention by the research team below:

1. Inform parents/guardians and children (over 9 years old) of their child's infection with toxocariasis and counseling to participate in treatment.
2. Counseling to participate in the treatment course: Explain clearly the intervention process, the benefits and possible side effects when participating in the treatment course. If they agree, the parent/guardian and the child (over 9 years old) will sign a consent form to participate in phase 2.
3. Distribute albedazol (Zentel) 200mg at school to guardians, dose 15mg/kg divided into 2 times/day, guide to take the medicine in full dose, at the right time after eating, taking full day 5
4. Advice on prevention of reinfection: feeding children cooked food, deworming dogs, handling dog feces, washing hands when touching soil, washing hands before eating, do not hold dogs/cats....
5. Instruct family members to monitor unwanted effects of albedazol (abdominal pain, nausea, urticaria, itching, allergic reactions...), if any, contact the research team's phone number for guidance and treatment according to the guidance of the Ministry of Health.
6. Schedule a follow-up visit after 1 month, clinical assessment.
7. Control medication compliance: daily, the research team will call parents to remind them to take the medicine, put the pill pack in the child's school bag to send back to the medical control agency. , and ask about the side effects of the drug or not.
8. Schedule a follow-up visit after 6 months from taking the drug, clinical assessment, blood collection as in the process of stage 1, repeat TPM, AST, ALT, Urea, Creatinine, IgE, ELISA. ,
9. Nurturing children. In case of suspected heart, lung, liver, eye damage, etc., we will refer you to Children's Hospital 2 for examination by specialty and not for intervention.

Standard operating procedures Examination procedure The research team coordinated with the school administration and the school health department to organize a visit at the school.

Examination of children is carried out by pediatricians of Pham Ngoc Thach University of Medicine with seniority, prestige, and practice certificates, undergraduate and postgraduate teaching jobs at Children's Hospital 2.

Procedures for taking blood samples, storing and transporting samples and handling accidents Sample Place of implementation: At the school of the child selected for the study. Test type: Complete blood count (TPTTBM), AST-ALT, Urea Creatinine, IgE, ELISA Performer: Pediatric nurse with seniority working at Children's Hospital 2, with good practice and professional certificates.

Blood volume: 4ml (divided into 3 specialized tubes: 0.5ml for BM; 1.5ml for urea-creatinine, AST-ALT, IgE; 2ml for ELISA) Storage and transportation Blood samples are stored at 4 - 8ºC in a dedicated shipping container and transported to Children's Hospital 2 laboratory 2 hours before the time of sampling according to the correct procedure Handling accidents Equip shockproof box and appropriate on-site first aid equipment, handle according to the protocol of the Ministry of Health, transfer the child to the nearest medical facility.

Procedure for performing the test Place of implementation: Laboratory of Children's Hospital 2 (hematology, biochemistry, microbiological diagnosis) Technique of ELISA test to find antibodies to Toxocariasis larvae. Test principles

* Microwells are coated with exocrine antigens of Toxocara larvae. During the first incubation with the patient's diluent serum, if any antibodies react with the antigen, they will bind to the antigen-coated wells. After washing off the remainder of the sample, add the conjugate enzyme.
* During the second incubation, the conjugate enzyme will bind to any antibodies present. After a second wash, a coloring agent (tetramethylbenzidine or TMB) is added. In the presence of the conjugate enzyme, peroxidase catalyzes the use of peroxide to turn the colorant blue. The blue color turns yellow after the addition of the stopping solution. Results are read visually or using an ELISA reader.

Sample collection and preparation Serum or plasma is stored at 2-8 0C for five days. Serum can be kept longer if stored at -20ºC for a long time. Do not freeze whole blood samples. Do not heat the sample and avoid freezing and thawing many times.

Read the results ELISA reader: reads zero with air. Set up a dual wavelength readout at 450/620-650 nm.

Positive: Absorbance reading is more than 0.3 OD units. Negative: Absorbance reading is less than 0.3 OD units. Information of the Toxocara ELISA Kit used for testing

* Test Toxocara IgG ELISA
* Kit name AccuDiag™ Toxocara IgG ELISA Kit
* Country of manufacture: America
* Method Enzyme-linked immunosorbent
* Skill Sandwich complex
* Detection threshold Qualifying: positive or negative
* Sample 5 L serum/plasma
* Test time ~ 20 minutes
* Expiry date 12 months from date of manufacture
* Specificity 93.3%
* Sensitivity 87.5%
* Circulation license number Number: 8362NK/BYT-TB-CT, March 9, 2018 of the Ministry of Health

Procedure for monitoring and taking care of children during treatment During the time the intervention group takes albedazol, the research team will coordinate with the school health department to monitor the children's clinical manifestations, call parents and guardians to assess unwanted effects of medication, reminders of treatment adherence, and preventive measures.

Procedure for recording side effects, adverse events, and adverse event handling

* Instruct family members to monitor unwanted effects of albedazol (abdominal pain, nausea, urticaria, itching, allergic reactions...), if any, contact the research team's phone number for advice. advice and guidance.
* Depending on the severity of the reaction, the research team will advise monitoring if the reaction is mild, or guide hospitalization for treatment and management according to the guidance of the Ministry of Health if the reaction is severe (Appendix 4). When determining that this reaction is caused by albedazol, the child's treatment costs will be covered from the project's funding (Section 11 Appendix 8)
* Record unwanted effects according to the ADR report form (Appendix 6) and send information to the National Center for Drug Information and Adverse Drug Reaction Monitoring (Hanoi University of Pharmacy:13- 15 Le Thanh Tong, Hoan Kiem District, Hanoi, email: di.pvcenter@gmail.com ).

Ethics This study was carried out through clinical examination, blood collection for routine tests and oral Albedazol intervention. We only conduct tests and drug interventions with the consent of the family and the school (signed the agreement through the consent form).

During the research, children are always monitored and evaluated for complications as well as side effects of drugs; If any, they will be consulted or treated according to the guidance of the Ministry of Health and the treatment costs will be covered from the project's budget.

This study was conducted with the approval of the Biomedical Research Ethics Council of Pham Ngoc Thach University of Medicine Ho Chi Minh City.

Funding: Department of Science and Technology of Ho Chi Minh City, Vietnam.

ELIGIBILITY:
Inclusion Criteria for phase 1 study:

* Pupils aged 3-15 years from Kindergarten to Secondary schools
* Agreement from parents with writen informed consent

Inclusion criteria for intervention:

* Children infected with toxocariasis may have symptoms and the ELISA test is positive for Toxocariasis larvae, with or without increased BCAT and IgE.

ELISA results according to the specified Kit and read according to optical densities (OD).

Cases of suspected heart, lung, liver, eye damage ... referred to Children's Hospital 2 for examination by specialty and not for intervention.

Exclusion Criteria:

* Children aged 3-15 years without writen informed consent from parents and themselves.
* Children infected with Toxocariasis larvae which are not common type.
* Children infected with Toxocariasis are suffering from acute diseases or other chronic diseases: Cardiovascular, hepatitis, kidney, stomach, mental, or suspected tumor...
* Children with a history of hypersensitivity to any ingredient in the treatment of Albendazole.
* Infected children do not have enough follow-up process before and after 1, 6 months of treatment.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 960 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Procedures Guidelines for diagnosis, treatment, and post-treatment follow-up of Toxocariasis larvae | 12 months
  After phase 1, we hope that we can draw a new procedure guideline for the diagnosis and treatment. And after this study is done, the new standard of guidelines for treatment of Toxocariasis infection can be applied for all children hospital in Vietnam.

SECONDARY OUTCOMES:
Seminars on treatment and follow-up after treatment of toxocariasis | 12 months
  After the phase 1 of the study, we can oganize the seminars based on the knowledge we have reviewed and will discuss about the treatment and follow-up to all the medical doctors who are interested in this topic.
Pet care consultation club, how to prevent toxocariasis | 12 months
  This club will invite the parents and anyone who care about taking care of animals such as dogs, cats at the family participate in this consultation club to provide information related to Toxocariasis infection and will educate them how to prevent infecting from Toxocariasis for children at home.
Publishing journal articles | 24 months
  Based on the reviewing the epidemiology and the situation about Toxocariasis in Vietnam, we can publish an article on it. After the phase 1 is done, we can publish the second article and after the phase 2 is done, we can publish the third one.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ha TV, Tang HK, Ngo BV, Le TPT, Le DH, Tran YML, Dang DKH, Vo TTN. Clinical and laboratory characteristics of Toxocara canis infection among children in Ho Chi Minh City, Vietnam. Trans R Soc Trop Med Hyg. 2025 Jan 3;119(1):27-32. doi: 10.1093/trstmh/trae057. PMID 39253804